CLINICAL TRIAL: NCT07098026
Title: Shenqi Fuwei Mixture Combined With Chemotherapy Neoadjuvant Therapy for Locally Advanced Gastric Cancer: A Multicenter Randomized Controlled Clinical Study
Brief Title: Shenqi Fuwei Mixture Combined With Chemotherapy Neoadjuvant Therapy for Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HNCH-2024KY81
Record Dates: First submitted 2025-06-15; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer, Adenocarcinoma
Keywords: locally advanced gastric cancer; perioperative; neoadjuvant chemotherapy; Shenqi Fuwei Mixture
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Multicenter, large-sample, randomized, double-blind, placebo-controlled clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, investigators, image assessors, and statistical analysts were blinded and emergency letters were set up to unblind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shenqi Fuwei Mixture (Experimental): Shenqi Fuwei Mixture
  Interventions: Drug: Shenqi Fuwei Mixture
- Shenqi Fuwei Mixture Placebo (Placebo Comparator): Shenqi Fuwei Mixture Placebo
  Interventions: Drug: Shenqi Fuwei Mixture Placebo

INTERVENTIONS:
Drug: Shenqi Fuwei Mixture — Shenqi Fuwei Mixture
  Arms: Shenqi Fuwei Mixture
Drug: Shenqi Fuwei Mixture Placebo — Shenqi Fuwei Mixture Placebo
  Arms: Shenqi Fuwei Mixture Placebo

SUMMARY:
The purpose of this clinical trial is to investigate whether the drug Shenqi Fuwei Mixture is effective for postoperative recurrence and metastasis of gastric cancer. Safety of Shenqi Fuwei Mixture will also be understood. It aims to answer the main questions:

* Shenqi Fuwei Mixture in perioperative combined with neoadjuvant chemotherapy to reduce the recurrence and metastasis of locally advanced gastric cancer after surgery?
* Shenqi Fuwei Mixture in the prevention and treatment of postoperative recurrence and metastasis of gastric cancer dominant population characteristics and efficacy mechanism?
* Exploratory excavation of TCM syndrome, multi-omics combined means to explore the advantages of Shenqi Fuwei Mixture on postoperative recurrence and metastasis of gastric cancer? The researchers will compare the drug Shenqi Fuwei Mixture with placebo (a substance that does not contain drugs and has a similar appearance) to see if the drug Shenqi Fuwei Mixture can prevent and treat recurrence and metastasis of gastric cancer after surgery.

Participants will:

* Take Shenqi Fuwei Mixture or placebo daily, synchronize with chemotherapy, or until tumor progression or intolerable toxicity
* Visits every 3 weeks for tests and tests
* Their survival status and adverse drug reactions were recorded

ELIGIBILITY:
Inclusion Criteria:

* Gastric or gastroesophageal junction adenocarcinoma confirmed by pathology or cytology;
* Resectable or potentially resectable gastric cancer with clinical stage of cT3-4aN + M0 or cT4bNxM0;
* Patients who are not allowed to receive previous anti-tumor therapy including chemotherapy radiotherapy immunotherapy or targeted therapy; Adequate organ function defined as follows: hematological ANC ≥ 1.5 * 10 ^ 9/L hemoglobin ≥ 9 g/dL platelets ≥ 80 * 10 ^ 9/L albumin ≥ 30 g/L serum bilirubin ≤ 1.5 × ULN AST and ALT ≤ 2.5 × ULN ALP ≤ 2.5 × ULN TBIL ≤ 1.5 × ULN renal serum creatinine < 1.5 × ULN.
* KPS ≥ 70 points;
* 18-75 years old male or female;
* Subjects voluntarily signed a written informed consent form.

Exclusion Criteria:

* Associated with distant metastasis;
* Patients with known hypersensitivity or metabolic disorder to fluorouracil or oxaliplatin or known hypersensitivity or intolerance to the study drug; Patients with primary malignant tumors at other sites. Subjects who were disease-free for 5 years or had a history of completely resected non-melanoma skin cancer or successfully treated carcinoma in situ were eligible;
* Gastrointestinal emergencies include: inability to swallow (complete or incomplete) gastrointestinal obstruction gastrointestinal bleeding and gastrointestinal perforation;
* Patients who are pregnant have neurological diseases or mental illness and mental and language disorders;
* Known uncontrolled angina pectoris arrhythmia congestive heart failure or myocardial infarction or a history of cardiac insufficiency within 6 months prior to study enrollment;
* Any concurrent disease or condition that may make the subject unsuitable for study participation or any serious medical condition that may interfere with the subject 's safety;
* Persons who are incapable (legally) or unsuitable for continuing study treatment for ethical/medical reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
EFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Event-Free Survival

SECONDARY OUTCOMES:
Surgical conversion rate | Binary classification variables were used to calculate the proportion of patients who could undergo surgery, whichever came first, assessed up to 60 months
OS | From date of randomization until the date of death from any cause, whichever came first, assessed up to 60 months
  Overall Survival
Tumor markers | "Baseline" or "3 week"
  CEA、CA724、CA199、CA125
DFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Disease-Free Survival
Infections and complications | Perioperative/Periprocedural
FACT-Ga Scale | "Baseline" or "At the begin of Cycle 1 (each cycle is 21 days)"
  Functional Assessment of Cancer Therapy--Gastric cancer Scale. minimum and maximum values: 0-100, and higher scores mean a better outcome.
Adverse events | At the end of Cycle 1 (each cycle is 21 days)
ESAS Scale | "Baseline" or "At the begin of Cycle 1 (each cycle is 21 days)"
  Edmonton Symptom Assessment Scale. minimum and maximum values: 0-100, and higher scores mean a better outcome.
MDASI-TCM Scale | "Baseline" or "At the begin of Cycle 1 (each cycle is 21 days)"
  M.D.Anderson Symptom Inventory Traditional Chinese Medicine Scale. minimum and maximum values: 0-100, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes